CLINICAL TRIAL: NCT06316063
Title: Hemodynamic Effects of Apnoeic Oxygenation With High-flow Nasal Oxygen in Adults Undergoing Laryngeal Surgery - a Randomised Study
Brief Title: Hemodynamic Effects of Apnoeic Oxygenation With High-flow Nasal Oxygen in Adults Undergoing Laryngeal Surgery
Acronym: CAPOX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Stockholm (Other Government)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2023-
Record Dates: First submitted 2024-03-12; First posted 2024-03-18 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2024-11

CONDITIONS: Laryngeal Disease
Keywords: Apnoeic oxygenation; Pulmonary hypertension; High-flow nasal oxygen; Right ventricular function
MeSH Terms: conditions — Laryngeal Diseases; Hypertension, Pulmonary | interventions — Respiration, Artificial

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Apnoeic oxygenation with High-flow nasal oxygen (Experimental): In the apnoeic oxygenation group the HFNO is used for pre-oxygenation,100 % O2, 40 L/min during 3 min. Thereafter, anaesthesia is induced by intravenous Propofol and Remifentanil. Rocuronium for full neuromuscular blockade is administered and a jaw thrust is used to keep an open airway. The airway will be kept patent throughout the procedure using a suspension laryngoscope, placed by the ENT surgeon. During apnoea oxygen will be increased to 70 L/min, 100% O2. Apnoea will be discontinued if any of the criteria SpO2 < 90%, PaCO2 >11 kPa, pH <7.15 or arrhythmias with haemodynamic effects occur.
  Interventions: Device: Apnoeic oxygenation with high-flow nasal oxygen
- Mechanical ventilation (Active Comparator): In the mechanical ventilation group pre-oxygenation is performed by a tight-fitting facemask, 100 % O2, for three minutes. After anaesthesia induction and full neuromuscular blockade, tracheal intubation is performed and mechanical ventilation is started.
  Interventions: Other: Mechanical ventilation

INTERVENTIONS:
Device: Apnoeic oxygenation with high-flow nasal oxygen — The subjects in the intervention group will be oxygenated with HFNO during the surgical procedure.
  Arms: Apnoeic oxygenation with High-flow nasal oxygen
Other: Mechanical ventilation — Study subjects in the comparator group will be tracheally intubated and mechanically ventilated
  Arms: Mechanical ventilation

SUMMARY:
During apnoeic oxygenation there is a continuous raise in carbon dioxide with subsequent respiratory acidosis. The hypercapnia and respiratory acidosis have several dose-related effects on both the systemic and the pulmonary circulation and the heart that ultimately, if unrecognised, can result in cardiovascular collapse and fatal arrhythmias. In our knowledge, no studies have investigated the haemodynamic effects of apnoeic oxygenation with HFNO.

The general purpose of this project is to investigate haemodynamic alternations during apnoeic oxygenation with HFNO compared to mechanical ventilation in relatively healthy patients under general anaesthesia during laryngeal surgery.

DETAILED DESCRIPTION:
This study aims to investigate and observe the circulatory effects in a patient undergoing apnoeic oxygenation with HFNO during shorter elective laryngeal surgery compared to mechanical ventilation. 20 patients scheduled for elective laryngeal surgery, eligible for apnoeic oxygenation at the Karolinska University Hospital, will be recruited. If eligible, the patient will receive oral and written study information by one of the investigators well in advance of the planned surgery. After a signed consent, the subject will be enrolled and randomised to either apnoeic oxygenation with HFNO or mechanical ventilation.

Patient characteristics such as age, sex, weight, height, ASA classification, other comorbidities and airway-related parameters will be documented. A preoperative transthoracic echocardiographic examination and routine perioperative monitoring, will be performed together with a 12-lead ECG. Preoperatively, an arterial catheter will be inserted in the radial artery and an arterial blood gas, measuring PaCO2, PaO2, pH, HCO3 and blood samples of stress markers including catecholamines and other cardiac biomarkers will be collected. The FloTrac system will be connected to the arterial catheter and baseline values will be registered. A peripheral venous catheter is placed prior to anaesthesia and the patient is placed supine.

In the apnoeic oxygenation group the HFNO nasal prongs (Optiflow, Fisher & Paykel Healthcare, Auckland, New Zealand) is placed in the nostrils and used for pre-oxygenation, 100 % O2, 40 L/min during 3 min. Thereafter, anaesthesia is induced by intravenous Propofol and Remifentanil administration. Rocuronium for full neuromuscular blockade is administered and a jaw thrust is used to keep an open airway. The start of apnoea is noted, defined as 1 minute after Rocuronium administration. The airway will be kept patent throughout the procedure using a suspension laryngoscope, placed by the ENT surgeon.

During apnoea the flow of oxygen is increased to 70 L/min, 100% O2. Apnoea will be discontinued if any of the criteria SpO2 < 90%, PaCO2 >11 kPa, pH <7.15 or arrhythmias with haemodynamic effects occur. In the mechanical ventilation group pre-oxygenation is performed by a tight-fitting facemask, 100 % O2, for three minutes. After anaesthesia induction using intravenous Propofol and Remifentanil and Rocuronium for full neuromuscular blockade, tracheal intubation is performed and mechanical ventilation is started. The start of apnoea is noted. The ventilator is set to PEEP 5 cmH2O, tidal volume (TV) 7 ml/kg ideal body weight, FiO2 0.4, and the respiratory frequency adjusted to reach a PaCO2 of 5,0 -5,3 kPa. Standard perioperative monitoring will be registered (peripheral oxygen saturation, heart rate and MAP). Arterial blood gases will be collected and ECG performed repeatedly. Data from the FloTrac system will be monitored throughout the procedure. Transthoracic echocardiography will be performed regularly. Blood samples to analyse stress markers including catecholamines and cardiac biomarkers will be collected at specific timepoints.

At the end of the procedure, any neuromuscular blockade is reversed by Sugammadex. The end of apnoea is defined as reoccurrence of spontaneous breathing or start of mask ventilation. In the mechanically ventilated group, subjects are extubated when awake and responsive.

After the procedure and when fully awake, the patient is transferred to the post-operative unit. The FloTrac monitoring will be continued during the postoperative period and the TTE, ECG evaluation, arterial blood gases, stress markers including catecholamines and cardiac biomarkers will be repeated during the post-operative period. Routine postoperative monitoring will be performed for a minimum of 60 minutes.

ELIGIBILITY:
Inclusion criteria

* Adult, ≥18 years old
* ASA 1-2
* BMI < 30
* Planned for elective laryngeal surgery

Exclusion criteria

* NYHA-class >1
* Pregnancy
* Severe gastric reflux
* Neuromuscular disease
* Any pulmonary disease
* Smokers or former smoker, last finished 6 months before inclusion
* Not capable of understanding study information and signing a written consent

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-03-25 (Actual); Primary Completion 2024-11-26 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Significant haemodynamic effects during apnoeic oxygenation with HFNO | 3 hours
  Significant haemodynamic effects such as significant increase in mPAP and/or new echocardiographic signs of right ventricular strain or failure compared to baseline, during and up to 2 hours after apnoeic oxygenation with HFNO or mechanical ventilation.

SECONDARY OUTCOMES:
Alterations in FloTrac derived central haemodynamic parameters | 3 hours
  Alterations in FloTrac derived central haemodynamic parameters such as MAP, SV, SVRI and CI, during and up to 2 hours after apnoeic oxygenation with HFNO or mechanical ventilation.
Alterations in Electrocardiogram | 3 hours
  Alterations in electrocardiogram during and up to 2 hours after apnoeic oxygenation with HFNO or mechanical ventilation.
Alterations in arterial carbon dioxide, oxygen and pH | 3 hours
  Alterations in arterial carbon dioxide, oxygen and pH during and up to 2 hours after apnoeic oxygenation with HFNO or mechanical ventilation.
Alterations in blood catecholamines and cardiac biomarkers | 3 hours
  Alterations in blood catecholamines and cardiac biomarkers during and up to 2 hours after apnoeic oxygenation with HFNO or mechanical ventilation.

CONTACTS AND LOCATIONS:
Overall Officials: Malin Jonsson Fagerlund, Principal Investigator — Region Stockholm
Locations (1):
- Karolinska Universitetssjukhuset Huddinge, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No